CLINICAL TRIAL: NCT05782127
Title: A Phase I/II, Open-label, Single Arm, Multicenter Dose-finding Study Assess the Safety and Preliminary Efficacy of Oral Azacitidine CC-486 (ONUREG) in Combination With Venetoclax (VENCLYXTO) in Previously Untreated Higher-risk Myelodysplastic Syndromes Ineligible for Allogenic Transplantation
Brief Title: Oral Azacitidine Combined With Venetoclax in Previously Untreated Higher-risk Myelodysplastic Syndromes
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Bristol-Myers Squibb (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-ONUVEN-MDS; 2022-000634-41 (EudraCT Number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Untreated Myelodysplastic Syndrome
Keywords: MDS; Oral Azacitidine; Venetoclax
MeSH Terms: interventions — venetoclax; cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Onureg + Venetoclax (Experimental): Onureg (CC-486, oral azacitidine) will be administered orally at 200 or 300 mg once daily for 7 or 14 consecutive days, beginning on Day 1 of repeated 28-day cycles.
  Venetoclax will be administered orally at 400 mg once daily for 14 consecutive days on days 1 to 14, beginning on Day 1 of repeated 28-day cycles.
  Patients will be treated up to 4 cycles and for a maximum of 24 cycles.
  Interventions: Drug: Onureg + Venetoclax

INTERVENTIONS:
Drug: Onureg + Venetoclax — Combination of Onureg and Venetoclax
  Other Names: CC-486 + ABT-199

SUMMARY:
This phase I/II open-label, dose-finding, multi-center study will assess safety and primary efficacy of Onureg and Venetoclax combination, to define the optimal biological dose and optimal treatment duration of Onureg to be used along with Venetoclax for further studies in previously untreated patients with higher-risk myelodysplastic syndromes (HR-MDS) not eligible to transplant.

DETAILED DESCRIPTION:
During phase I, three dose features of Onureg will be tested in combination with a fixed dose of Venetoclax to define the optimal biological dose for phase II.

The phase II will assess safety and primary efficacy of Onureg and Venetoclax combination, to define the optimal biological dose and optimal treatment duration of Onureg to be used along with Venetoclax for further studies in previously untreated patients with HR-MDS not eligible to transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand and voluntarily sign and date an ICF indicating the investigational nature of the study, approved by an independent EC/IRB, prior to the initiation of any screening or study-specific procedures.
2. Age ≥ 18 years at the date of signing the ICF.
3. Diagnosis of MDS according to the 2016 WHO classification (13) (Appendix 1), with presence of < 20% bone marrow blasts per bone marrow aspirate at screening, confirmed by local investigator with HR-MDS, based on the revised International Prognostic Scoring System (IPSS-R) >3 (intermediate, high or very high) (14) (Appendix 2) and a blast percentage of 5 or more.
4. Previously untreated HR-MDS: no prior therapy for MDS with any hypomethylating agents (azacitidine or decitabine), chemotherapy, allo-Hematopoietic Stem Cell Transplantation (HSCT) or experimental agent. All other treatments are not considered prior therapy.
5. Not immediately eligible for allo-HSCT or intensive chemotherapy at the time of screening due to individual clinical factors such as age, comorbidities and performance status, donor availability.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Total white blood cell (WBC) count ≤ 10 G/L; Treatment with hydroxyurea is permitted to lower the WBC to reach this inclusion criterion and will be stopped at least 48 hours before treatment initiation.
8. Adequate liver functions as demonstrated by:

   * Serum alanine transaminase (ALT) < 3.0 × upper limit of normal [ULN];
   * Serum aspartate transaminase (AST) < 3.0 × ULN;
   * Serum total bilirubin ≤ 2.0 × ULN (except in the setting of isolated Gilbert syndrome, where participants may only be included with total bilirubin ≤ 3.0 x ULN)
9. Adequate renal function with calculated creatinine clearance ≥ 40 mL/min/1.73 m² (estimation based on Modification of Diet in Renal Disease (MDRD) formula or CKD-EPI, by local laboratory).
10. Participant is able to communicate with the investigator, and has the ability to comply with the requirements of the study procedures, available for regular blood sampling, study related assessments, including bone marrow aspirates and appropriate clinical management at the treating institution for the duration of the study.
11. Females of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months). FCBP must agree to undergo medically supervised pregnancy test prior to starting study drug, during the course of the study, and after end of study therapy:

    * Have one negative pregnancy test as verified by the Investigator prior to starting study therapy. The first pregnancy test will be performed at screening (within 3 days prior to first study drug administration), and a negative urinary test before starting all subsequent cycles. This applies even if the participant practices true abstinence from heterosexual contact or agree to use, and be able to comply with highly effective contraception without interruption, 28 days prior to starting investigational product, during the study therapy (including dose interruptions), and for 6 months after last dose of Onureg, or at least 1 month after the last dose of venetoclax, whichever is later or longer if required by local regulations.
    * Female patients are either post-menopausal, free from menses for > 2 years, surgically sterilized or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agree to abstain from becoming pregnant throughout the study, starting with Visit 1. Females of reproductive potential as well as fertile men and their partners who are female of reproductive potential must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the study and for 6 months (females and males) following the last dose of treatment.
12. Male participants must practice true abstinence (which must be reviewed on a monthly basis) or agree to use an adequate method of contraception for the duration of the study. Men should be advised not to father a child while receiving treatment and for 3 months post study. Men must agree to learn about the procedures for preservation of sperm before starting treatment.

Exclusion Criteria:

1. Previous treatment for MDS, any approved or investigational antineoplastic agents or radiotherapy.
2. Previous diagnosis of:

   * MDS evolving from a pre-existing myeloproliferative neoplasm (MPN)
   * MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN.
3. Participant has an active, uncontrolled systemic fungal, bacterial, or viral infection. The participant should be afebrile and off antibiotics for at least 72 hours and off antifungals for 7 days. In the case of prior SARS-CoV-2 infection, symptoms must have completely resolved and based on Investigator assessment in consultation with the Medical Monitor, there are no sequelae that would place the patient at a higher risk of receiving investigational treatment.
4. History of clinically significant medical conditions, laboratory abnormality, psychiatric illness or any other reason that the investigator determines would interfere with the subject's participation in this study, would make the subject an unsuitable candidate to receive study drug or predisposes the participant to high risk of noncompliance with the protocol.
5. History of active malignancy within the past year prior to screening, with the exception of:

   * Adequately treated carcinoma in situ of the uterine cervix
   * Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
   * Asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy.

   Patients with ongoing horomonotherapy could be included.
6. Participant has received strong or moderate CYP3A inhibitors or inducers or p-gp inhibitors within 7 days prior to initiation of study treatment with prolonged treatment required without therapeutic alternatives. Azols are the only exception and may be permitted after cycle 1 at investigator's discretion and will result in venetoclax dose reduction.
7. Consumption of grapefruit products, Seville oranges or starfruit within 3 days prior to first dose of venetoclax.
8. Received live attenuated vaccines prior to initiation of study treatment.
9. History of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months.
10. Conditions that could interfere with drug absorption including short gut syndrome, dysphagia, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
11. Participant has uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 100 mmHg) or has not been stable for at least 1 month prior to treatment.
12. Significant active cardiac disease within the previous 6 months prior to signing the ICF, including:

    * New York Heart Association (NYHA) Class III or IV congestive heart failure
    * Unstable angina or angina requiring surgical or medical intervention
    * Significant cardiac arrhythmia
    * And/or myocardial infarction
13. Participant is a pregnant or lactating female.
14. Participant has known or suspected to have hypersensitivity to any of the components of the assigned study treatments.
15. Positive test result(s) for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Subjects with serologic evidence of prior vaccination to hepatitis B virus (i.e., hepatitis B surface antigen [HBsAg] negative, anti-hepatitis B surface [HBs] antibody positive and anti-hepatitis B core [HBc] antibody negative) may participate.
16. Absence of social security affiliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | at day 28 of cycle 1
  Dose-limiting toxicities according to CTCAE (common terminology criteria for adverses events) 5.0 occurring within the first cycle of treatment
Overall response | at day 28 of cycle 1
  Overall response measured after the first cycle of treatment according to modified IWG-MDS (International Working Group-Myelodysplastic Syndromes) 2006

SECONDARY OUTCOMES:
Best response | after 6 cycles of treatment (each cycle is 28 days)
  Best response evaluated according to the modified IWG-MDS 2006 and IWG-HR-MDS 2023 criteria
Hematological improvement | at end of treatment (an average of 4 years)
  Hematological improvement (erythroid, neutrophil and platelet improvement) according to IWG-MDS 2006 and IWG-HR-MDS 2023
Time to response | at end of treatment (an average of 4 years)
  Time from onset of treatment to date of achievement of any response according to the modified IWG-MDS 2006 criteria
Duration of response | at end of study (an average of 5 years)
  Time interval between the first date of achievement of any response according to the modified IWG-MDS 2006 criteria to relapse
Progression to acute myeloid leukemia (AML) | at end of treatment (an average of 4 years)
  Rate of transformation to AML
Time to next treatment | at end of study (an average of 5 years)
  Time from onset of trial treatment to onset of subsequent therapy
Survival | at end of study (an average of 5 years)
  Determination of overall survival rate, event-free survival rate, progression-free survival rate
Transfusion independence | at end of study (an average of 5 years)
  Rate of red blood cells and platelets transfusion independance for transfusion-dependent patients at baseline
Duration of transfusion independence | at end of study (an average of 5 years)
  Time interval between the achievement of transfusion independence and relapse with need of transfusion
Identification and grading of adverse events | at end of treatment (an average of 4 years)
  Toxicity profile of study treatment including identification and grading of adverse events based on NCI CTCAE version 5, cytopenia duration, life-threatening or fatal cytopenias rate, unscheduled hospitalization rate, infectious complications rate, red blood cells and platelets transfusions needs
Patient-reported outcomes according to FACIT-AN | at end of treatment (an average of 4 years)
  Patient-reported outcomes according to Functional Assessment of Chronic Illness Therapy - anemia (FACIT-An) version 4 (Score range: 0-188), evaluation of of change in QoL from baseline
Early mortality | at day 28
  Determination of early mortality rate at day 28
Patient-reported outcomes according to EQ-5D-5L | at end of treatment (an average of 4 years)
  Patient-reported outcomes according to 5-level EuroQol-5D (EQ-5D-5L) (Scale numbered from 0 to 100), evaluation of change in QoL from baseline
Patient-reported outcomes according to PGIC | at end of treatment (an average of 4 years)
  Patient-reported outcomes according to Patient global impression of change (PGIC) form, evaluation of change in QoL from baseline
Patient-reported outcomes according to PGIS | at end of treatment (an average of 4 years)
  Patient-reported outcomes according to Patient global impression of severity (PGIS) form, evaluation of change in QoL from baseline

OTHER OUTCOMES:
Exploratory endpoints by NGS | end of study (an average of 5 years)
  Determination of minimal Residual Disease (MRD) by Next Generation Sequencing (NGS) and dynamics of molecular alterations associated with MDS
MRD response rate | end of study (an average of 5 years)
  Determination of MRD negative NGS rate

CONTACTS AND LOCATIONS:
Overall Officials: Colombe SAILLARD, MD, Principal Investigator — Institut Paoli-Calmettes; Norbert VEY, MD/PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (25):
- France (25):
  - CHU d'Amiens Picardie - Site sud, Amiens
  - CHU d'Angers, Angers
  - Hôpital Avicenne, Bobigny
  - Hôpital privé Sévigné, Cesson-Sévigné
  - CH Annecy Genevois, Épagny
  - CHU de Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - CH Lyon sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHI Mont-de-Marsan, Mont-de-Marsan
  - CHU Saint Eloi, Montpellier
  - CHU Hôtel Dieu, Nantes
  - Hôpital Archet 1, Nice
  - CHU Nîmes - Institut de Cancérologie du Gard, Nîmes
  - Hôpital Saint Louis, Paris
  - Hôpital Cochin, Paris
  - CHU de Haut-Lévèque, Pessac
  - CHU de Poitiers, Poitiers
  - Centre Henri Becquerel, Rouen
  - IUCT Oncopole, Toulouse
  - CHU de Tours - Hôpital Bretonneau, Tours
  - CH Valence, Valence
  - Hôpital Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No